CLINICAL TRIAL: NCT03654742
Title: Intracapsular vs Extracapsular Tonsillectomy. A Comparison of Treatment Methods of Recurrent and Chronic Tonsillitis in Adults: a Prospective Single-blinded Randomised Study
Brief Title: Intracapsular Tonsillectomy in Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Jaakko Piitulainen, Consultant, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: T211/2018
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Tonsil Disease; Tonsillitis; Tonsillitis Acute; Tonsillitis Chronic
Keywords: tonsil surgery; tonsillectomy; intracapsular; microdebrider; coblation; extracapsular; electrosurgery; electrocautery; adults
MeSH Terms: conditions — Tonsillitis; Hyperthermia | interventions — Tonsillectomy

STUDY DESIGN:
Intervention Model Description: prospective, single-blinded, randomised, controlled
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients are masked with numbers and patient records not shown to the outcomes assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ECTE/Electrosurgery (Active Comparator): Extracapsular tonsillectomy (ECTE) with monopolar electrosurgery
  Interventions: Procedure: tonsillectomy
- ICTE/Microdebrider (Experimental): Intracapsular tonsillectomy (ICTE) with microdebrider
  Interventions: Procedure: tonsillectomy
- ICTE/Coblator (Experimental): Intrapsular tonsillectomy (ICTE) with coblator
  Interventions: Procedure: tonsillectomy

INTERVENTIONS:
Procedure: tonsillectomy — removal of tonsil tissue as described in the study arms
  Other Names: tonsil removal; tonsil surgery

SUMMARY:
Comparing the classical extracapsular tonsillectomy (TE) performed with electrosurgery to intracapsular approaches (SIPT) by coblation or microdebrider. The patient group is adults with recurrent or chronic tonsillitis

DETAILED DESCRIPTION:
Extracapsular tonsillectomy (TE) with monopolar electrosurgery is the most commonly used approach in adult tonsil surgery in Turku University Central Hospital, Finland.

In our study setting we are comparing intracapsular tonsillectomy (subtotal/intracapsular/partial tonsillectomy (SIPT) ) as the intervention group with extracapsular tonsillectomy as the control group.

SIPT is done with either coblation or microdebrider and TE with monopolar electrosurgery.

Indications for surgery are recurrent tonsillitis or chronic tonsillitis. The patient group is adults (16-65 years)

Safety, efficiency and cost-effectiveness are monitored in a prospective, patient-blinded and randomised study setting.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-65 years
* Planned tonsil surgery with informed consent
* Recurrent or chronic tonsillitis

Exclusion Criteria:

* Less than 1 month old, drained quinsy
* Acute "hot phase" tonsillitis
* Previous palatine tonsil surgery
* Suspicion or confirmation of malignancy
* High dose analgesics consumption
* Current CPAP-device usage for treatment of OSAS
* Untreated gastro-esophageal reflux disease
* Anticoagulative medication
* Any condition of hemophilia
* Pregnancy, lactation
* Current or positive history of malignant disease (if still active follow-up)

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Post-operative recovery | 21 days
  Pain post-operatively after discharge as self-reported pain intensity over the past day. Each day is scored with the modified Brief Pain Inventory and recovery is achieved when pain score reaches preset values. Recovery speed defined as pain VAS-score 3 or less at rest; or pain VAS-score 5 or less without regular analgesics use. Daily questionnaire used: Brief Pain Inventory.

SECONDARY OUTCOMES:
Analgesics use | 21 days
  Need for analgesics postoperatively during 21 days. Measured as number of naprometin tablets/ day and the number of tramadol-paracetamol combination tablets/day.
Post-operative bleeding | 21 days
  Bleeding post-operatively at the ward or at any point during 21 days. Measured as 1-4 (1= bleeding, stopped spontaneously, no contact with staff; 2: Contact with ER, bleeding stopped without intervention; 3: Bleeding, needed intervention (packing, topical adrenalin, electrosurgical hemostasis; 4: Needed OR-time, blood transfusion, ward days
Life Quality | 6 months
  Quality of life as defined by the questionnaires: Tonsillectomy Outcome Inventory 14 "TOI-14" preoperatively and 6 months after operation;
Residual tonsil tissue | 6 months
  Residual tonsil measured right after surgery is completed and at 6 months follow-up.
Revision surgery | 5 years
  The need of revision surgery after tonsillectomy, recorded with questionnaire: Nordic Tonsil Surgery Register
Throat problems | 5 years
  Throat problems as described by the Nordic Tonsil Surgery Register at different time points postoperatively
Life quality | 6 months
  Quality of life as defined by the questionnaires: Glasgow Benefit Inventory "GBI" at 6 months after operation.

CONTACTS AND LOCATIONS:
Overall Officials: Jussi Jero, Professor, Study Director — Turku University Hospital
Locations (1):
- TYKS Korvaklinikka, Turku, Finland

IPD SHARING:
Plan to Share IPD: Yes
All data relevant to the study are included in the article or uploaded as supplementary information.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available with the publication of the article

REFERENCES:
- [Background] Piitulainen JM, Uusitalo T, Sjoblom HM, Ivaska LE, Jegoroff H, Kauko T, Kokki H, Kyto E, Mansikka I, Ylikoski J, Jero J. Intracapsular tonsillectomy in the treatment of recurrent and chronic tonsillitis in adults: a protocol of a prospective, single-blinded, randomised study with a 5-year follow-up (the FINITE trial). BMJ Open. 2022 Sep 14;12(9):e062722. doi: 10.1136/bmjopen-2022-062722. PMID 36104143